CLINICAL TRIAL: NCT04367051
Title: Withdrawal of Spironolactone Treatment for Heart Failure With Improved Left Ventricular Ejection Fractraction: an Open-label Randomized Controlled Pilot Study (With-HF Trial)
Brief Title: Pilot Study on Withdrawal of Spironolactone Among Heart Failure With Improved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang Eun Lee, professor of medicine, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_2020_0613
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Withdrawal group (Experimental): Spironolactone will be discontinued in patients who were receiving optimal medical therapy including angiotensin-converting enzyme or angiotensin receptor blocker or angiotensin receptor neprilysin, beta-blocker, and spironolactone.
  Interventions: Drug: Withdrawal of Spironolactone
- Continuation group (Active Comparator): Spironolactone will be continued during the study period with other medical therapy in combination.
  Interventions: Drug: Continuation of spironolactone

INTERVENTIONS:
Drug: Withdrawal of Spironolactone — Other recommended medications for heart failure than spironolactone will be continued for withdrawal group.
  Arms: Withdrawal group
Drug: Continuation of spironolactone — Specific dose of spironolactone for continuation group is on each physician's discretion with acceptable range of 12.5 mg - 50 mg once or twice daily.
  Arms: Continuation group

SUMMARY:
The study is a randomized controlled pilot trial to evaluate whether withdrawal of spironolactone is safe and associated with re-deterioration of left ventricular function in patients with heart failure with improved ejection fraction. The aim of current trial is to test the hypothesis that withdrawal of spironolactone would not be associated with relapse of significant clinical deterioration of left ventricular systolic function.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of providing informed consent and agrees to follow the study protocol and schedule of clinical follow-up
* Age between 19 and 80 years old
* Prior diagnosis of heart failure with reduced left ventricular ejection fraction (LV EF ≤ 35%) and on medical therapy including spironolactone combined with angiotensin-converting enzyme or angiotensin receptor blocker or antiotensin receptior neprilysin blocker, beta-blocker.
* LV EF ≥ 50% documented with echocardiography performed within a month
* Documented result of BNP or NT-proBNP level within a month

Exclusion Criteria:

* Dyspnea ≥ New York Heart Association (NYHA) functional class III
* Patients who need to discontinue spironolactone owing to prior adverse event
* Primary valvular heart disease with at least moderate degree
* Estimated glomerular filtration rate less than 30 mL/min per 1.73 m2
* Uncontrolled hypertension defined as blood pressure more than 140/90 mmHg
* Presence of other clinical reason to continue spironolactone such as myocardial infarction, primary aldosteronism, and liver cirrhosis
* Hyperkalemia defined as serum potassium level less than 3.5 mmol per liter
* Pregnant and/or lactating women
* Life expectancy less than a year
* Patients who are not suitable to enrollment by investigator's discretion

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change of left ventricular ejection fraction | 6 month
  Proportion of patients with change of left ventricular ejection fraction declining more than 10%

SECONDARY OUTCOMES:
Numerical change of left ventricular ejection fraction | 6 month
  Comparison as continuous variable
Change of serum level on B-type natriuretic peptide or N-terminal pro-brain natriuretic peptide | 6 months
  Each serum level transformed with a log value and comparing with baseline level
Change of serum level of biomarkers (e.g. soluble ST-2, galectin-3) | 6 months
  Serum biomarkers such as soluble ST-2, galectin-3 are checked and compared with baseline value for prediction of decreased left ventricular ejection fraction
Rates of death, re-hospitalization or visit on emergency department for heart failure | 6 months
  Adverse clinical events
results of each outcomes during extended follow-up period | 2 years
  change of echocardiographic parameters, clinical events, natriuretic peptide

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hyun J, Lee SA, Lee SE, Hong JA, Kim MS, Kim JJ. Withdrawal of Spironolactone for Heart Failure With Improved Ejection Fraction: An Open-Label, Pilot, Randomized Controlled Trial (With-HF Trial). Korean Circ J. 2025 Dec;55(12):1077-1089. doi: 10.4070/kcj.2025.0052. Epub 2025 Jul 8. PMID 40736394